CLINICAL TRIAL: NCT00325728
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of 8 Week Treatment of Rozerem 8 mg (QHS) in Sleep Disturbed, Mild to Moderately Severe Alzheimer's Disease Subjects
Brief Title: Efficacy and Safety of Ramelteon in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-061; U1111-1115-1644 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Sleep Initiation and Maintenance Disorder; Drug Therapy; Alzheimer disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alzheimer Disease | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8mg, tablets, orally, once nightly for up to 8 weeks.
  Other Names: TAK-375; Rozerem
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo matching tablets, orally, once nightly for up to 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of ramelteon, once daily (QD), in subjects with mild to moderate Alzheimer's Disease and sleep disturbance

DETAILED DESCRIPTION:
Epidemiological data for 2005 show that an estimated 4.2 million people in the US suffer from Alzheimer's disease, often necessitating caregiver assistance, which can in many cases progress to institutionalization. Subjects with Alzheimer's disease dementia frequently experience disturbed sleep patterns characterized by insufficient nocturnal sleep and excessive daytime napping, which has been associated with both cognitive and behavioral pathology such as impaired daytime functioning, agitation, and nocturnal wandering.

Although the causality of sleep disturbances in Alzheimer's disease remains unclear; some research suggests that the fragmented sleep and associated behavioral disturbances could be related to the degeneration of the serotonergic and noradrenergic innervation of suprachiasmatic nucleus andsubsequent disruption in melatonin secretion patterns. Additionally, research suggests that melatonin levels are decreased in patients with Alzheimer's disease

In the United States, ramelteon is marketed for the treatment of insomnia characterized by difficulty with sleep onset and is under global development for the treatment of transient, chronic insomnia and circadian rhythm sleep disorders. It is believed that ramelteon works by binding melatonin to MT1/MT2 receptors in the suprachiasmatic nucleus which inhibits firing of specific neurons, which is thought to attenuate the alerting signal and allows the homeostatic mechanism to express itself and promote sleep.

Study participation is anticipated to be about 11 weeks (approximately 3 months).

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of dementia of the Alzheimer's type (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised) or probable Alzheimer's disease by National Institute of Neurological and Communicative Disorders and Stroke/the Alzheimer's Disease and Related
* Disorders Association criteria.
* Female subjects must be post-menopausal.
* Stable residence with no planned move during the entire investigation period.
* Residing in the same residence with a responsible spouse, family member, or a professional caregiver who is present during the night who would agree to assume the role of the principal caregiver for the duration of the protocol period.
* Able to ingest oral medication and participate in all scheduled evaluations.
* Clinical laboratory evaluations (including clinical chemistry, hematology, and urinalysis) within the reference range as tested by the designated laboratory unless the results are deemed not clinically significant by the investigator or sponsor.
* Treatment medications for any non-excluded medications or concurrent medical conditions are stable for 30 days prior to the screening visit and medication(s) can in the investigator's judgment, remain stable throughout the duration of the study.
* Mini-Mental State Examination score of 8 to 28, inclusive.
* History of greater than or equal to 2 sleep disorder behaviors, occurring at least once weekly over the two weeks before screening.
* Actigraphy evidence shows a nighttime total sleep time of less than 7 hours per night based on at least 4 out of 7 nights of complete actigraphy data collected over the single-blind, placebo run-in period.
* Habitual bedtime of between 8 PM and 12 AM.

Exclusion Criteria

* Non-ambulatory, wheel chair bound or confined to bed and is without a consistent caregiver who is present during the night who could function as the primary caregiver.
* Caregiver is deemed by the investigator to be unreliable to supervise the wearing of the actigraphy, to complete the sleep log, to administer medication at the proper time, to bring the subject to the scheduled visits or to answer questions regarding the subject's condition or medication use.
* Lacks a mobile upper extremity to which to attach an actigraphy.
* Currently participating or has participated in another clinical study within the past 30 days.
* Demonstrates an unwillingness to abstain from caffeine after 2:00 PM for the duration of the clinical trial participation.
* Demonstrates an unwillingness to comply with the maximum limit of two alcoholic drinks per day and only one alcoholic drink after 6:00 PM for the duration of the protocol.
* Uses tobacco products or any other products during nightly awakenings that may interfere with the sleep wake cycle.
* History of drug abuse or tests positive for the presence of illicit drugs.
* Donated more than 400 mL of blood within the 90 days preceding the beginning of the study.
* Diastolic blood pressure greater than 95 mm Hg or a systolic pressure of greater than 160 mm Hg.
* Body mass index of greater than 36.
* Alanine transaminase level of greater than two times the upper limit of normal, active liver disease, jaundice or any clinically significant abnormal laboratory findings as determined by the investigator.
* History of a hypersensitivity or allergies to Ramelteon or melatonin.
* History of contraindications as noted in the Ramelteon label
* History of significant stroke or vascular dementia.
* History of severe renal dysfunction or disease.
* History of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.)
* Any clinically significant movement disorder including but not limited to: akinesia, periodic limb movement disorder, restless leg syndrome, epilepsy, uncontrolled Parkinson's disease, or severe benign prostatic hyperplasia, cardiac asthma, chronic obstructive pulmonary disease.
* Rapid eye movement behavior disorder or sleep apnea.
* Any pain syndrome affecting sleep.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Fluvoxamine
  * Melatonin
  * Rifampicin

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-03-21 (Actual); Primary Completion 2007-08-01 (Actual); Study Completion 2007-08-20 (Actual)

PRIMARY OUTCOMES:
Mean Nighttime Total Sleep Time as determined by actigraphy. | Week 1

SECONDARY OUTCOMES:
Change from Baseline in Nighttime Total Sleep Time | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in Nighttime Wake After Sleep Onset per Actigraphy | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in Nighttime Number Of Awakenings per Actigraphy | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in Daytime Total Sleep Time | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in the ratio of Daytime Total Sleep Time to Nighttime Total Sleep Time. | Weeks 2, 4, 6, and 8 or Final Visit
Change from Baseline in Sleep Efficiency. | Weeks 2, 4, 6, and 8 or Final Visit
Percentage of subjects who experience Increase in Nighttime Total Sleep Time of 30 minutes. | Weeks 2, 4, 6, and 8 or Final Visit
Number of Daytime Naps. | Weeks 2, 4, 6, and 8 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research and Development
Locations (72):
- United States (72):
  - Alabaster, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Fresno, California
  - Irvine, California
  - Los Angeles, California
  - National City, California
  - Oxnard, California
  - San Diego, California
  - San Francisco, California
  - Darien, Connecticut
  - Waterbury, Connecticut
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Brooksville, Florida
  - Deerfield Beach, Florida
  - Fort Myers, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - Orange City, Florida
  - Pompano Beach, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Boston, Massachusetts
  - West Yarmouth, Massachusetts
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Dover, New Hampshire
  - Piscataway, New Jersey
  - Princeton, New Jersey
  - Stratford, New Jersey
  - Toms River, New Jersey
  - Whiting, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - New Hyde Park, New York
  - New York, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Havertown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Moon Township, Pennsylvania
  - Philadelphia, Pennsylvania
  - Beaufort, South Carolina
  - Greer, South Carolina
  - North Charleston, South Carolina
  - Bellaire, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Bennington, Vermont
  - Burlington, Vermont
  - Middleton, Wisconsin

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI